CLINICAL TRIAL: NCT02385383
Title: An Intravenous Iron Based Protocol for Optimizing Haemoglobin in Anaemic Patients Prior to Fast-track Hip and Knee Arthroplasty - An Observational Follow up Study
Brief Title: An Intravenous Iron Based Protocol for Preoperative Anaemia in Hip and Knee Surgery - An Observational Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Hvidovre University Hospital (Other); Bispebjerg Hospital (Other); Gentofte Hospital (Unknown); Vejle Sygehus (Unknown); Regionshospitalet Viborg, Skive (Other); Farsø Sygehus (Unknown)
Responsible Party: Principal Investigator, Oeivind Jans, M.D., Ph.D., Rigshospitalet, Denmark
Other Study IDs: RH-4074-OJ4
Record Dates: First submitted 2015-02-16; First posted 2015-03-11 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Anemia; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Patient Blood Management; Preoperative anemia; IV Iron
MeSH Terms: conditions — Anemia | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with preoperative anemia following treatment protocol: Patients with preoperative anemia according to the WHO definition and treated with a protocol of Iitravenous iron prior to surgery
  Interventions: Drug: Iron-III Isomaltoside 1000
- Patients with preoperative anemia - Historical control: Cohort of preoperative anemic patients from the Lundbeckcentre Database. Serving as a historical control
  Interventions: Other: Standard Care

INTERVENTIONS:
Drug: Iron-III Isomaltoside 1000 — Protocol for optimizing preoperative Hb using IV Iron-III Isomaltoside 1000
  Other Names: Monofer
  Groups: Patients with preoperative anemia following treatment protocol
Other: Standard Care — Standard Care in a historical control cohort
  Groups: Patients with preoperative anemia - Historical control

SUMMARY:
This observational study follows a cohort of patients scheduled for elective hip- or knee surgery but has preoperative anemia and are treated with Intravenous (IV) iron prior to surgery according to a recently introduced standardized treatment protocol at 6 high-volume surgical centres.

DETAILED DESCRIPTION:
Patients presenting with preoperative anaemia prior to hip and knee arthroplasty has a high risk of receiving allogeneic blood transfusion and anaemia has been associated with increased postoperative morbidity and mortality. While IV-iron administration may raise Hb prior to surgery, existing guidelines for addressing and treating preoperative anaemia is not widely implemented for patients scheduled for elective total joint arthroplasty (TJA) in Denmark. In addition, causes of preoperative anaemia and the efficacy of preoperative IV-iron administration has not been sufficiently evaluated in elective TJA.

This is a observational follow-up study among 6 Danish high volume surgical centres that has recently introduced a standardized anaemia screening and treatment protocol for patients with preoperative anaemia scheduled for total hip- or knee arthroplasty.

Patients with iron deficiency anaemia or anaemia of chronic inflammation receive infusion of IV-iron (Monofer) 4 weeks prior to surgery as a part of the standard operating procedure on the department.

The aim of this follow up study is to evaluate changes in Haemoglobin concentration, transfusion rate and postoperative morbidity in this cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Scheduled for elective primary hip- or knee arthroplasty
* Preoperative hemoglobin < 13 g/dl (males) or < 12 g/dl (females)
* Included in the departments treatment protocol for preoperative anemia

Exclusion Criteria:

* Cronic transfusion need
* Not able to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective hip or knee arthroplasty presenting with preoperative anemia.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Transfusion Rate | From date of admission to date of discharge (up to 30 days)
  Blood transfusion (yes/no) during the entire hospital stay

SECONDARY OUTCOMES:
Classification of preoperative anemia | 4 weeks prior to surgery (baseline)
Change in hemoglobin concentration | From date of preoperative blood sampling (baseline) to date of admission (Up to 4 weeks)
  The change in Hb from the time of preoperative blood sampling to Hb sampled on the date of admission
No. of red blood cell units administered per patient | From date of admission to date of discharge (up to 30 days)
  No of blood units administered during the entire hospital stay
Length of Hospital stay | From date of admission to Date of discharge (up to 30 days)
Postoperative complications and readmissions | From date of surgery up to 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Oeivind Jans, M.D., Ph.D., Principal Investigator — Rigshospitalet, Denmark
Locations (6):
- Denmark (6):
  - Bisbebjerg Hospital, Dept. of orthopedic surgery, Copenhagen NV
  - Farsø Sygehus, Farsø
  - Gentofte Hospital, Dept. of orthopedic surgery, Hellerup
  - Hvidovre Hospital, Department of orthopaedic surgery, Hvidovre
  - Vejle Sygehus, Dept. of orthopedic surgery, Vejle
  - Viborg Sygehus, Dept. of orthopedic surgery, Viborg